CLINICAL TRIAL: NCT01489046
Title: A Phase IIb Randomized, Controlled, Partially Blinded Clinical Trial to Investigate Safety, Efficacy and Dose-response of BMS-986001 in Treatment-naive HIV-1-infected Subjects, Followed by an Open-label Period on the Recommended Dose
Brief Title: Safety, Efficacy and Dose-response Study of BMS-986001 in Subjects With HIV-1 Infection Who Are Treatment-naive
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI467-003; 2011-003329-89 (EudraCT Number)
Record Dates: First submitted 2011-12-07; First posted 2011-12-09 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — BMS-986001; efavirenz; Lamivudine; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1: BMS-986001 (100 mg) + Placebo + Efavirenz + Lamivudine (Experimental)
  Interventions: Drug: BMS-986001; Drug: Placebo matching with BMS-986001; Drug: Efavirenz; Drug: Lamivudine
- Arm 2: BMS-986001 (200 mg) + Placebo + Efavirenz + Lamivudine (Experimental)
  Interventions: Drug: BMS-986001; Drug: Placebo matching with BMS-986001; Drug: Efavirenz; Drug: Lamivudine
- Arm 3: BMS-986001 (400 mg) + Efavirenz + Lamivudine (Experimental)
  Interventions: Drug: BMS-986001; Drug: Efavirenz; Drug: Lamivudine
- Arm 4: Tenofovir (300 mg) + Efavirenz + Lamivudine (Experimental)
  Interventions: Drug: Efavirenz; Drug: Lamivudine; Drug: Tenofovir

INTERVENTIONS:
Drug: BMS-986001 — Capsules, Oral, 100 mg, Once daily, At least 48 weeks
  Arms: Arm 1: BMS-986001 (100 mg) + Placebo + Efavirenz + Lamivudine
Drug: BMS-986001 — Capsules, Oral, 200 mg, Once daily, At least 48 weeks
  Arms: Arm 2: BMS-986001 (200 mg) + Placebo + Efavirenz + Lamivudine
Drug: BMS-986001 — Capsules, Oral, 400 mg, Once daily, At least 48 weeks
  Arms: Arm 3: BMS-986001 (400 mg) + Efavirenz + Lamivudine
Drug: Placebo matching with BMS-986001 — Capsules, Oral, 0 mg, Once daily, At least 48 weeks
  Arms: Arm 1: BMS-986001 (100 mg) + Placebo + Efavirenz + Lamivudine; Arm 2: BMS-986001 (200 mg) + Placebo + Efavirenz + Lamivudine
Drug: Efavirenz — Tablets, Oral, 600 mg, Once daily, Entire Treatment Phase
  Other Names: Sustiva®
Drug: Lamivudine — Tablets, Oral, 300 mg, Once daily, Entire Treatment Phase
  Other Names: Epivir®
Drug: Tenofovir — Tablets, Oral, 300 mg, Once daily, Entire Treatment Phase
  Other Names: Viread®
  Arms: Arm 4: Tenofovir (300 mg) + Efavirenz + Lamivudine

SUMMARY:
The purpose of this study is to identify at least one dose of BMS-986001 which is safe, well tolerated, and efficacious when combined with Efavirenz (EFV) + Lamivudine (3TC) for treatment-naive Human Immunodeficiency Virus 1 (HIV-1) infected subjects

DETAILED DESCRIPTION:
Double Blind through Week 24. Partially Blind (to subjects, caregivers, Investigators) through Week 48.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, (or minimum age as determined by local regulatory or as legal requirements dictate, whichever is higher)
* Plasma HIV-1 RNA > 5000 copies/mL
* Antiretroviral treatment-naive; defined as no current or previous exposure to > 1 week of an antiretroviral drug
* CD4+ T-cell count > 200 cells/mm3

Exclusion Criteria:

* Resistance to any of the study medications [Tenofovir Disoproxil Fumarate(TDF), Efavirenz (EFV), Lamivudine (3TC)] or to HIV Protease Inhibitors (PIs)
* Contraindications to any of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2011-02; Primary Completion 2013-03 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with plasma HIV-1 RNA < 50 c/mL as measured by polymerase chain reaction (PCR) analyses | Week 24
Safety as measured by numbers of subjects with Serious Adverse Events (SAEs) and numbers of subjects with Adverse Events (AEs) leading to discontinuations | Week 24

SECONDARY OUTCOMES:
Proportion of subjects with plasma HIV-1 RNA < 50 c/mL as measured by PCR analyses | Weeks 48 and 96
Safety as measured by numbers of subjects with SAEs and numbers of subjects with AEs leading to discontinuation | Weeks 48 and 96
Changes from baseline in CD4+ T-cell counts | Weeks 24, 48, and 96
Numbers of subjects with virologic failure who exhibit genotypic substitutions in viral Ribonucleic acid (RNA) | Weeks 24, 48, and 96
Maximum observed concentration (Cmax) of BMS-986001 when co-administered with EFV and 3TC | Week 24
Time of maximum observed concentration (Tmax) of BMS-986001 when co-administered with EFV and 3TC | Week 24
Trough plasma concentration at 24 h post observed dose (Cmin) of BMS-986001 when co-administered with EFV and 3TC | Week 24
Trough plasma concentration pre-dose (C0) of BMS-986001 when co-administered with EFV and 3TC | Week 24
Area under the concentration-time curve in one dosing interval [AUC(0-24)] of BMS-986001 when co-administered with EFV and 3TC | Week 24
Average steady-state plasma concentration (Css,avg) of BMS-986001 when co-administered with EFV and 3TC | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (47):
- United States (18):
  - Uc Davis Medical Center, Sacramento, California
  - Orlando Immunology Center, Orlando, Florida
  - Triple O Medical Services, P.A., West Palm Beach, Florida
  - Aids Research Consortium Of Atlanta, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Local Institution, Washingtondc, Maryland
  - Clinic 42 And International Travel Clinic, Minneapolis, Minnesota
  - University At Buffalo, Buffalo, New York
  - Local Institution, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Local Institution, Charlotte, North Carolina
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Local Institution, Columbia, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - St. Hope Foundation, Bellaire, Texas
  - North Texas Infectious Disease Consultants, Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Therapeutic Concepts, P.A., Houston, Texas
- Local Institution, Ciudad de Buenos Aires, Buenos Aires, Argentina
- Australia (3):
  - Local Institution, Darlinghurst, New South Wales
  - Local Institution, Liverpool, New South Wales
  - Local Institution, Melbourne, Victoria
- Canada (2):
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Montreal, Quebec
- Local Institution, Santiago, Santiago Metropolitan, Chile
- Local Institution, Bogota, Cundinamarca, Colombia
- Local Institution, Lyon, France
- Local Institution, Budapest, Hungary
- Local Institution, Mexico City, Mexico City, Mexico
- Peru (4):
  - Local Institution, Barranco, Lima region
  - Local Institution, San Martín de Porres, Lima region
  - Local Institution, Cercado, Lima
  - Local Institution, Iquitos, Loreto
- South Africa (8):
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Soweto, Gauteng
  - Local Institution, Dundee, KwaZulu-Natal
  - Local Institution, Cape Town, Western Cape
  - Local Institution, Cape Town
  - Local Institution, Durban
  - Local Institution, Durban KZN
- Spain (3):
  - Local Institution, Badalona
  - Local Institution, Barcelona
  - Local Institution, Madrid
- Thailand (3):
  - Local Institution, Bangkok
  - Local Institution, Khon Kaen
  - Local Institution, Nontaburi

REFERENCES:
- [Derived] Gupta SK, McComsey GA, Lombaard J, Echevarria J, Orrell C, Avihingsanon A, Osiyemi O, Santoscoy M, Ray N, Stock DA, Joshi SR, Hanna GJ, Lataillade M. Efficacy, safety, bone and metabolic effects of HIV nucleoside reverse transcriptase inhibitor BMS-986001 (AI467003): a phase 2b randomised, controlled, partly blinded trial. Lancet HIV. 2016 Jan;3(1):e13-22. doi: 10.1016/S2352-3018(15)00231-3. Epub 2015 Dec 12. PMID 26762988
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx